CLINICAL TRIAL: NCT07082985
Title: Effects of Maca Supplementation on Badminton-specific Exercise Performance: Indicators of Exercise-Induced Fatigue and Oxidative Stress
Brief Title: Effects of Maca Supplementation on Badminton-specific Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Jung-Piao Tsao, Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CMUH112-REC2-148
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Athletes
Keywords: Black maca; Fatigue; Badminton
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: The study recruited twelve badminton athletes aged between 18 and 26 years, all of whom engage in regular physical training. Participants were crossed over for Maca or placebo supplements, which could be ended in two days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Containing edible yellow No. 4, edible yellow No. 5, sucrose, silica, talc, oxidized starch, gelatin, magnesium stearate, and palm wax.
  Interventions: Other: Placebo (Placebo trial); Other: Maca (Maca trial)
- Maca (Experimental): Each capsule containing 400 mg of Maca
  Interventions: Other: Placebo (Placebo trial); Other: Maca (Maca trial)

INTERVENTIONS:
Other: Placebo (Placebo trial) — The Placebo capsule supplement was taken for 14 days (4 capsules per day)
Other: Maca (Maca trial) — The Maca capsule supplement was taken for 14 days, with a daily dosage of 1600 mg of Maca (equivalent to 4 capsules per day, each containing 400 mg of Maca).

SUMMARY:
This study aims to investigate whether a 14-day short-term supplementation of Maca can effectively mitigate oxidative stress and fatigue induced by badminton competition.

DETAILED DESCRIPTION:
Maca possesses antioxidant and anti-fatigue properties, which may have potential positive effects on athletic performance. This study integrates Maca's physiological characteristics with the sport-specific demands of badminton to examine its impact on athletic performance. The experiment is designed as a single-blind, crossover trial involving 12 participants, each undergoing two trials: a placebo trial and a Maca supplementation trial, with a supplementation period of 14 days for both conditions.

On the test day, participants will be provided with a meal adjusted according to their body weight and will orally consume either Maca or a placebo capsule. After a one-hour rest period, they will perform a simulated badminton match. At the end of each game, participants will complete a 30-second cycling anaerobic power test, followed by a 1-minute and 30-second rest before starting the next game.

Finally, participants will undergo an aerobic capacity assessment through a badminton-specific progressive endurance test, which will continue until exhaustion. Blood samples will be collected both before and after the simulated badminton match for analysis of oxidative stress markers, including malondialdehyde (MDA) and superoxide dismutase (SOD), as well as fatigue markers, such as blood urea nitrogen (BUN) and creatine kinase (CK). Additionally, the total duration of the badminton-specific progressive endurance test will be recorded.

Furthermore, to assess participants' psychological states, the Profile of Mood States (POMS) questionnaire will be administered after both the simulated badminton match and the badminton-specific progressive endurance test.

ELIGIBILITY:
Inclusion Criteria:

* Badminton athletes aged between 18 and 26 years.
* Each with at least three years of playing experience and a regular exercise routine.

Exclusion Criteria:

* Have smoking and drinking habits.
* People who feel unwell due to other reasons during the experiment.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Badminton specific endurance test | Including for 2 days in both crossover trials (which lasts around 35 days).
  The research assistant will mark four points on the ground in a Y-shape configuration, with each target point positioned 3 meters away from the central point. The participant begins at the central point (P0). The participant must move to the upper-right Marker 1 (P1), touch the marker with the racket, and immediately return to P0. Next, the participant proceeds to Marker 2 (P2), touches it with the racket, and returns to P0. Then, the participant moves backward to Marker 3 (P3), and performs a badminton-specific turning jump along the central line to simulate a rear-court shot scenario, before returning again to P0. This entire sequence constitutes one round. The next round begins immediately after the previous one ends. This test is based on the average time of approximately 210 seconds reported by Wonish et al. (2003) for completing the test. The number of Y-shaped rounds completed within this total time is recorded as the participant's endurance performance.
Assessment of the profile of mood state (POMS) | Including for 2 days in both crossover trials (which lasts around 35 days).
  POMS brief was chosen for this study to evaluate the mood of individuals. After the "Badminton stimulation test" and "Badminton specific endurance test", participants completed the form, and their responses were analyzed using simple statistics. The results were shown in six dimensions, one positive: (1) vigor; and five negatives: (2) tension, (3) depression, (4) anger, (5) fatigue and (6) confusion.
Clinical Biochemistry of antioxidant and antifatigue biomarkers | Including for 2 days in both crossover trials (which lasts around 35 days).
  Blood sample were collected at two time points (before and after the badminton stimulation test). According to the manufacturer's instructions, Malondialdehyde (MDA) levels were measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit. Superoxide Dismutase (SOD) activity was determined using a commercial SOD activity assay kit, with absorbance analyzed via enzyme immunoassay. A commercial Uric Acid (UA) detection kit was used, and absorbance at 520 nm was measured using an automated enzyme immunoassay analyzer. For Creatine Kinase (CK), blood samples were collected and centrifuged at 1000 g for 20 minutes, with 0.5 mL of serum used for analysis. Absorbance was measured using an automated analyzer
30-second Wingate Test | Including for 2 days in both crossover trials (which lasts around 35 days).
  First, participants performed a 5-minute warm-up on a stationary 894E cycle ergometer with adjustable resistance at a low workload (50 W). Following the warm-up, resistance was set based on body weight (kg × 0.075), and participants completed three bouts of maximal effort sprints, each lasting 5 seconds. Between each sprint, participants pedaled at 50 W for 45 seconds as active recovery. During the test, strong verbal encouragement was provided by the staff to ensure maximal effort. For the main test, participants began pedaling at a cadence of 60 rpm. A verbal countdown (3, 2, 1) was given at an audible volume, and upon hearing the whistle, participants were instructed to immediately pedal with maximal speed and power for 30 seconds. The total and mean power output accumulated during the 30-second anaerobic performance test were recorded as indicators of anaerobic capacity.

SECONDARY OUTCOMES:
Badminton stimulation test | Including for 2 days in both crossover trials (which lasts around 35 days).
  The simulated badminton matches in this trial followed the most recent international competition rules established by the Badminton World Federation (BWF) in 2006, which adopt the "3 × 21 rally point scoring system." Participants were matched with opponents of similar skill levels based on a comprehensive assessment of their previous badminton performance (e.g., rankings, match footage review). The same opponent was used in both trials (Maca supplementation and placebo conditions). During the official test, each participant competed in a three-game singles, where the first player to reach 21 points wins the game. If the score reaches 20-20, the game continues until one player leads by two consecutive points or reaches 30 points first. All other match rules, such as scoring, fouls, and court changes, adhered strictly to official BWF regulations.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Piao Tsao, Study Chair — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No